CLINICAL TRIAL: NCT06000722
Title: The Generation of Expert Consensus-based Clinical Guidelines for the Use of Sodium-glucose Co-transporter 2 (SGLT2) Inhibitors in Patients With Diabetic Foot Ulcer Disease: a Delphi Study
Brief Title: SGLT-i Use in Diabetic Foot Ulcer Disease
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 40318
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare practitioners: Participants who are trained healthcare practitioners involved in the care of patients with current or previous diabetic foot ulcer disease
  Interventions: Other: eDelphi method

INTERVENTIONS:
Other: eDelphi method — This is a Delphi technique-based study using a purposive sample of convenience. Consensus development methods will be used to generate clinical guidelines, endorsed by key clinical groups, on the use of SGLT2i's in patients with diabetic foot ulcer disease, including acknowledgement of specific scenarios or patient characteristics that may influence these guidelines.

SUMMARY:
Background: People with diabetes and either current or previous diabetic foot ulcer disease (DFUD) are at very high risk for adverse cardiovascular events including heart attacks and strokes. Sodium-glucose co-transporter 2 (SGLT2) inhibitors are a class of medications that have shown to be very effective in reducing heart disease and event risk. However, one recent study found that SGLT2i's may increase minor amputation risk in those with DFUD, though this finding has not been replicated in other similar studies. However, as a result, there has been limited further investigation into this issue and as such the use of SGLT2i's in those with DFUD remains a contentious issue, despite their potential for significantly reducing cardiovascular disease risk in this population.

In the absence of further randomised controlled trials investigating the use of SGLT2is in these populations, there is a need for clinical guidelines advising on their use based on expert clinical consensus, including specific criteria or scenarios in which they should or should not be used. The Delphi methodology is an iterative survey technique that uses expert opinion from various relevant backgrounds and experiences to generate a consensus based upon various statements and/or scenarios.

Aim: The aim of this study is to use the Delphi technique to generate expert consensus-based clinical guidelines on the use of SGLT2i's in those with diabetes and DFUD.

Methods: This is a Delphi technique-based study using a purposive sample of convenience. Consensus development methods will be used to generate clinical guidelines, endorsed by key clinical groups, on the use of SGLT2i's in patients with diabetic foot ulcer disease, including acknowledgement of specific scenarios or patient characteristics that may influence these guidelines.

The consensus group will consist of n=20 healthcare practitioners, including GPs, secondary care diabetologists, foot care specialists, cardiologists and pharmacists in order to ensure a breadth of expertise and input. Two rounds of the Delphi consensus process will take place, in order to iteratively develop the consensus-based clinical guidelines. This process is expected to take 4-6 months. The analysis will be on-going throughout the study and completed within 3 months of the last questionnaire round of the Delphi process.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are trained healthcare practitioners involved in the care of patients with current or previous diabetic foot ulcer disease

Exclusion Criteria:

* Potential participants who do not give informed consent. Potential participants who will not be able to participate in both rounds of the Delphi process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the Delphi study will consist of n=20 healthcare practitioners and will be recruited from a convenience sample, and representing a range of specialties and clinical backgrounds.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Delphi Round 1 | 3 weeks
  Each participant will provided with the clinical statements regarding the use of SGLT2i's in patients with diabetic foot ulcer disease, and sent the link to an online questionnaire. Within the first questionnaire round the participants will be asked to rate these statements i.e. strongly agree, agree, uncertain (probably agree), uncertain (probably disagree), disagree, strongly disagree. Participants will be given three weeks to complete this questionnaire, and will be sent reminder emails during this time. This will establish priorities amongst the statements listed. As a result of completing round one, areas of disagreement and agreement will be identified and a level of consensus will begin to form.
Delphi Round 2 | 3 weeks
  The second round of the questionnaire will consist of a summary of the items and ratings from the previous round. Participants will be asked to revise his/her judgments or to specify why they wish to remain outside of the consensus. This round gives the Delphi participants an opportunity to make further clarifications of both the information & their judgment of the relative importance of the items. Round 2 will be initiated 1 month after the completion of round 1. If consensus is not reached on the majority of statements following round 2, and third and final round may be added in order to reach consensus.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester, United Kingdom